CLINICAL TRIAL: NCT01731665
Title: Epidemiology of Inflammatory Bowel Disease in the Songpa-Kangdong District, Seoul, Korea.
Status: Recruiting | Type: Observational
Sponsor: Asan Medical Center (Other)
Collaborators: Kyung Hee University Hospital at Gangdong (Other); Seoul National University Hospital (Other); Seoul National University Bundang Hospital (Other); Samsung Medical Center (Other); Konkuk University Medical Center (Other); National Police Hospital (Other Government); Seoul Veterans Hospital (Other); hansol hospital (Unknown); Kangdong Seoul Clinic (Other); Jamsil Seoul Surgical Clinic (Unknown); Song Do Colorectal Hospital (Unknown); Yang Hospital (Other); Daehang Hospital (Other); Kangdong Sacred Heart Hospital (Other)
Responsible Party: Principal Investigator, Suk-Kyun Yang, Professor, Asan Medical Center
Other Study IDs: 2012-0634
Record Dates: First submitted 2012-11-18; First posted 2012-11-22 (Estimated); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Crohn's Disease; Ulcerative Colitis; Epidemiology; Korea
Keywords: Crohn's disease; ulcerative colitis; epidemiology; Korea
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- The Songpa-Kangdong cohort of IBD: Incident cases of IBD in the Songpa-Kangdong district, a well-defined administrative area in Seoul, the capital of Korea, beginning in 1986, when the first patient with IBD was diagnosed, until 2017. For the prevalent cases, the inhabitants with IBD at Dec 31, 2007 in the Songpa-Kangdong district are included.

SUMMARY:
The purpose of this study is to evaluate the incidence, prevalence, clinical characteristics and prognosis of Crohn's disease and ulcerative colitis over time in a district of Seoul, Korea.

DETAILED DESCRIPTION:
Inflammatory bowel disease (IBD), which is comprised of Crohn's disease (CD) and ulcerative colitis (UC) is a chronic inflammatory disease of gut with uncertain etiopathogenesis. According to our previous study (Yang, et al. Inflamm Bowel Dis 2008; 14: 542-549), the incidence and prevalence of IBD in Korea are still low compared with those in Western countries, but are rapidly increasing. However, the long-term trends of epidemiology of CD and UC together with their characteristics and prognosis in Korea are uncertain yet. The investigators therefore aim to elucidate the incidence and prevalence of CD and UC over a 30-year period, from 1986 to 2017, in the Songpa-Kangdong district of Seoul, Korea. In addition, the investigators also aim to reveal the clinical features at the time of diagnosis of IBD, long-term evolution of disease and prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Definite cases of CD and UC

Patients are diagnosed with CD if they meet at least 2 of the following criteria:

1. clinical history of abdominal pain, weight loss, malaise, diarrhea, and/or rectal bleeding
2. endoscopic findings of mucosal cobblestoning, linear ulceration, skip areas, or perianal disease
3. radiologic findings of stricture, fistula, mucosal cobblestoning, or ulceration
4. macroscopic appearance of bowel wall induration, mesenteric lymphadenopathy, and "creeping fat" at laparotomy
5. pathologic findings of transmural inflammation and/or epithelioid granulomas

Only patients who meet these criteria for at least 2 months are included.

Patients are diagnosed with UC only if all 3 of the following criteria are present

1. a typical history of diarrhea or blood and pus or both in the stool for longer than 4 weeks
2. a typical sigmoidoscopic or colonoscopic picture with diffusely granular, friable, or ulcerated mucosa without rectal sparing or skip lesions or radiological signs of characteristic continuous granular or ulcerated mucosa
3. characteristic histopathological signs of inflammation on biopsy

Exclusion Criteria:

* IBD unclassified
* Ethnic groups other than Korean

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study is performed in the Songpa-Kangdong district, a well-defined administrative area in Seoul, the capital of Korea, beginning in 1986, when the first patient with IBD was diagnosed, until 2017. The population of the study area was racially and ethnically homogeneous and was relatively stable in number.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2012-12 (Actual); Primary Completion 2029-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Incidence rate and prevalence rate of IBD | 1986-2017 (up to 31 years)
  1. Annual incidence rate of Crohn's disease and ulcerative colitis
  2. Prevalence rate of Crohn's disease and ulcerative colitis as of Dec 31, 2017.

SECONDARY OUTCOMES:
Clinical features of patients with IBD | 1986-2017 (up to 31 years)
  1. Clinical characteristics of patients newly diagnosed with Crohn's disease or ulcerative colitis: gender, presenting symptoms, duration between symptoms to diagnosis, and phenotypes, etc.
  2. Clinical course of patients newly diagnosed with Crohn's disease or ulcerative colitis: development of complications (strictures, perforations), intestinal resection rate, hospitalization rate, mortality, and pregnancies and their outcomes
  3. Treatment modalities of IBD and their trends: use of medication (5-ASA, corticosteroids, immunomodulators, and biologic agents, etc.)

CONTACTS AND LOCATIONS:
Overall Officials: Suk-Kyun Yang, M.D., Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yang SK, Yun S, Kim JH, Park JY, Kim HY, Kim YH, Chang DK, Kim JS, Song IS, Park JB, Park ER, Kim KJ, Moon G, Yang SH. Epidemiology of inflammatory bowel disease in the Songpa-Kangdong district, Seoul, Korea, 1986-2005: a KASID study. Inflamm Bowel Dis. 2008 Apr;14(4):542-9. doi: 10.1002/ibd.20310. PMID 17941073
- [Background] Yang SK, Hong WS, Min YI, Kim HY, Yoo JY, Rhee PL, Rhee JC, Chang DK, Song IS, Jung SA, Park EB, Yoo HM, Lee DK, Kim YK. Incidence and prevalence of ulcerative colitis in the Songpa-Kangdong District, Seoul, Korea, 1986-1997. J Gastroenterol Hepatol. 2000 Sep;15(9):1037-42. doi: 10.1046/j.1440-1746.2000.02252.x. PMID 11059934